CLINICAL TRIAL: NCT02812628
Title: Randomized Clinical Trial of Conventional Laparoscopic Abdominoperineal Resection (APR) Versus Laparoscopic APR With Transabdominal Individualized Levator Transection for Low Rectal Cancer
Brief Title: Conventional Laparoscopic APR Versus Laparoscopic APR With Transabdominal Individualized Levator Transection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Bo Feng, Assistent professor of surgery, Ruijin Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MISC-APR
Record Dates: First submitted 2016-06-10; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Rectal Cancer
Keywords: laparoscopic surgery; abdominoperineal resection; rectal cancer; individualized surgery; levator muscle
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional LAPR (Active Comparator): Patients undergoing conventional laparoscopic abdominoperineal resection (LAPR).
  Interventions: Procedure: LAPR
- LAPR-TILT (Experimental): Patients undergoing LAPR with transabdominal individualized levator transection (TILT).
  Interventions: Procedure: LAPR-TILT

INTERVENTIONS:
Procedure: LAPR — Patients undergoing conventional LAPR, the common surgical procedure to treat low rectal cancer ≤5m from anal verge.
  Arms: Conventional LAPR
Procedure: LAPR-TILT — Patients undergoing LAPR-TILT, a modified APR procedure that is supposed to be safer and less invasive as compared to the LAPR.
  Arms: LAPR-TILT

SUMMARY:
This study is designed to compare the short-term and long-term benefits between conventional laparoscopic abdominoperineal resection (APR) and laparoscopic APR with transabdominal individualized levator transection (TILT).

DETAILED DESCRIPTION:
In the field of surgical treatment for low rectal cancer, the traditional APR is trapped by the so-called "surgical waist" and associated oncological problems, whereas the spread of extra-levator abdominoperineal resection (ELAPR) is still hindered by its high risk of wound complications and neurovascular injuries. Owing to the advancement of laparoscopic techniques, the investigators developed a laparoscopic APR with TILT procedure. During the procedure, a controlled incision of levators into the ischiorectal fat was performed transabdominally under direct vision; the meeting plane is therefore lowered and the perineal dissection is simplified without changing body position. This technique offers individualized transection of levator muscles, minimizes the risk of wound complications and prevents surgical waist to ensure oncological safety. This clinical trial is designed to evaluate the short-term and long-term benefits of this modified procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as having rectal cancer ≤5cm from anal verge by colonoscopy.
2. Patients undergoing elective, radial surgery with no distant metastasis.
3. Patients with Body Mass Index (BMI) between 18-30kg/m2.
4. Patients who agree to undergo standard adjuvant treatment after surgery.
5. Patients who have fully understood the aim of the trial and have signed the written informed consent.

Exclusion Criteria:

1. Patients with distant metastasis, tumor infiltrating to adjacent organs, or recurrent tumors.
2. Patients undergoing emergent surgery.
3. Pregnant patients.
4. Patients with tumors other than rectal tumor.
5. Patients with severe comorbid diseases which preclude surgery.
6. Patients in bad conditions and do not ameliorate before surgery.
7. Patients undergoing other procedures to treat rectal cancer, eg. L-Dixon, L-Hartmann or Parks surgery.
8. Patients who refuse to accept standard adjuvant surgery.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Estimated)
Dates: Start 2012-12; Primary Completion 2020-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
3-year local recurrence | 3 years post operation

SECONDARY OUTCOMES:
3-year overall survival | 3 years post operation
3-year disease-free survival | 3 years post operation

OTHER OUTCOMES:
Operative time for perineal dissection | 1 month post operation
Numbers of days to remove the urinary catheter after surgery | 1 month post operation
Circumferential Resection Margin (+) rate | 1 month post operation
  circumferential resection margin positive rate
Perforation rate | 1 month post operation
  intraoperative perforation rate

CONTACTS AND LOCATIONS:
Overall Officials: Bo Feng, Ph.D, Principal Investigator — Ruijin Hospital
Locations (1):
- Ruijin Hospital affiliated to Shanghai Jiaotong University school of medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided